CLINICAL TRIAL: NCT03736993
Title: Towards Better Therapy for Resectable Lung Cancer: Metabolomics Predict Therapy Response
Brief Title: Metabolomics Predict Therapy Response
Acronym: PROLUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Prof. dr. Michiel Thomeer, Head of department of respiratory medicine, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PROLUNG001
Record Dates: First submitted 2018-08-17; First posted 2018-11-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: NSCLC, Stage IIIA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional blood sampling (Other): non-small cell lung cancer (NSCLC)
  Interventions: Other: Additional blood sampling

INTERVENTIONS:
Other: Additional blood sampling — Establish predictive markers for early disease progression after complete surgical resection in patients with stage I to IIIA NSCLC.

SUMMARY:
Complete resection is the mainstay of treatment for stage I-IIIA resectable non-small cell lung cancer (NSCLC). However rates of recurrence of disease are high, with five-year survival rates ranging between 73% (stage IA) and 24% (stage IIIA). Therefore, a prognostic biological marker that stratifies between NSCLC patients whom surgery cures versus patients in whom surgery would be futile due to early disease relapse after surgery is eagerly awaited.

The primary objective of this prospective study is to establish a prognostic marker of early disease progression after complete surgical resection in patients with stages I to IIIA NSCLC. For this purpose the investigator will compare the metabolic profile with disease progression or death within one year after complete surgical resection to the patients with a progression free survival. Furthermore the investigator will evaluate the changes in the metabolic profile after surgery and if changes in this metabolic profile over time can predict disease recurrence before it becomes clinically apparent.

DETAILED DESCRIPTION:
Introduction: Precision medicine relies on validated biomarkers that can accurately classify patients by their probable disease risk, prognosis and/or response to treatment. Metabolomics is particularly promising for biomarker development because altered metabolism is considered a hallmark of cancer. The measurement of the metabolomic plasma profile is cheap (+-50 EUR) and fast (+-17 min), with a high information throughput on a per sample base.

Rationale: Complete resection is the mainstay of treatment for stage I-IIIA resectable non-small cell lung cancer (NSCLC). However rates of recurrence of disease are high, with five-year survival rates ranging between 73% (stage IA) and 24% (stage IIIA). Therefore, a prognostic biological marker that stratifies between NSCLC patients whom surgery cures versus patients in whom surgery would be futile due to early disease relapse after surgery is eagerly awaited.

Study objective: The primary study hypothesis is that the metabolic plasma profile is a predictive marker of early disease progression after complete surgical resection in patients with pathological stages I to IIIA NSCLC. The secondary study hypothesis is that the level of dissimilarity between the metabolic profile before surgery and the metabolic profile after surgery, is a predictor for disease recurrence (in which the extreme case would be, that a normalization of the metabolic profile to the profile of a healthy person, is indicative of a good prognosis).

Study design: Prospective, interventional design

Study population: Stage I-IIIA NSCLC patients who will undergo complete surgical resection willing to provide a written informed consent.

Number of patients: 200 patients with stage I-IIIA NSCLC who will undergo thoracic surgery with a curative intent will be included.

Main study parameters/endpoints: Recurrence free survival, overall survival, metabolic phenotype, presence or absence of hot-spot mutations in tested proto-oncogenes and tumor suppressor genes in circulating tumor DNA (ctDNA) in blood plasma, the tumor tissue and possibly positive lymph nodes, 43 items of the EORTC quality of life questionnaire C30 and LC13.

Nature and extent of the burden and risks associated with participation: Subjects will be asked to give consent to take 10-30 ml of blood at several moments throughout the disease course and in follow-up. Furthermore, the participants need to give their permission to use the resected tumor/lymph node tissue for genetic testing. Clinical parameters will be pooled in a database in a confidential way.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a stage I-IIIA NSCLC tumor, eligible to undergo surgery
2. Signed written informed consent

Exclusion Criteria:

1. No fasting starting from 22:00 h the day prior to blood sampling
2. Medication intake in the morning of the blood sampling
3. Non-controlled diabetes
4. History of cancer during the past 5 years
5. Treatment for cancer during the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The metabolic profile in plasma measured by Nuclear Magnetic Resonance (NMR) | baseline
  The metabolic profile in plasma measured by Nuclear Magnetic Resonance (NMR) spectroscopy predicts disease disease recurrence within one year after surgical resection.

SECONDARY OUTCOMES:
Change in the metabolic profile in plasma measured by Nuclear Magnetic Resonance (NMR) | screening, day 1, week 1, week 4, week 6, week 12, week 52
  The degree of change in the metabolic profile in plasma before and after surgery correlates with the risk for early disease recurrence.
Change in ctDNA mutations in plasma | day 1, week 12, week 52
  The degree of change in ctDNA mutations in plasma before and after surgery correlates with the risk for early disease recurrence.
Correlation between presence or absence Hotspot mutations and the metabolic profile in plasma | day 1, week 12, week 52
  A specific metabolic profile in plasma measured by Nuclear Magnetic Resonance (NMR) spectroscopy correlates with the presence of absence of certain ctDNA mutations in plasma
Metabolic profile of the primary tumor | day 1
  The metabolic profile of the primary tumor correlates with the metabolic profile in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Thomeer, prof. dr., Principal Investigator — Hasselt University; Elien Derveaux, drs., Study Chair — Hasselt University; Liesbet Mesotten, prof. dr., Study Chair — Hasselt University; peter Adriaensens, prof. dr., Study Chair — Hasselt University
Locations (4):
- Belgium (4):
  - OLV ziekenhuis Aalst, Aalst
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: Undecided
still no plan for, but open for sharing after discussion with participating groups

REFERENCES:
- [Background] Louis E, Cantrelle FX, Mesotten L, Reekmans G, Bervoets L, Vanhove K, Thomeer M, Lippens G, Adriaensens P. Metabolic phenotyping of human plasma by 1 H-NMR at high and medium magnetic field strengths: a case study for lung cancer. Magn Reson Chem. 2017 Aug;55(8):706-713. doi: 10.1002/mrc.4577. Epub 2017 Feb 27. PMID 28061019
- [Background] Beger RD, Dunn W, Schmidt MA, Gross SS, Kirwan JA, Cascante M, Brennan L, Wishart DS, Oresic M, Hankemeier T, Broadhurst DI, Lane AN, Suhre K, Kastenmuller G, Sumner SJ, Thiele I, Fiehn O, Kaddurah-Daouk R; for "Precision Medicine and Pharmacometabolomics Task Group"-Metabolomics Society Initiative. Metabolomics enables precision medicine: "A White Paper, Community Perspective". Metabolomics. 2016;12(10):149. doi: 10.1007/s11306-016-1094-6. Epub 2016 Sep 2. PMID 27642271
- [Background] Beger RD. A review of applications of metabolomics in cancer. Metabolites. 2013 Jul 5;3(3):552-74. doi: 10.3390/metabo3030552. PMID 24958139
- [Result] Louis E, Adriaensens P, Guedens W, Bigirumurame T, Baeten K, Vanhove K, Vandeurzen K, Darquennes K, Vansteenkiste J, Dooms C, Shkedy Z, Mesotten L, Thomeer M. Detection of Lung Cancer through Metabolic Changes Measured in Blood Plasma. J Thorac Oncol. 2016 Apr;11(4):516-23. doi: 10.1016/j.jtho.2016.01.011. Epub 2016 Feb 29. PMID 26949046
- [Result] Louis E, Adriaensens P, Guedens W, Vanhove K, Vandeurzen K, Darquennes K, Vansteenkiste J, Dooms C, de Jonge E, Thomeer M, Mesotten L. Metabolic phenotyping of human blood plasma: a powerful tool to discriminate between cancer types? Ann Oncol. 2016 Jan;27(1):178-84. doi: 10.1093/annonc/mdv499. Epub 2015 Oct 20. PMID 26487580